CLINICAL TRIAL: NCT02043002
Title: Early Changes in 18F-fluorodeoxyglucose Positron Emissions Tomography (18F-FDG-PET/CT) Scan as Predictors of Clinical Outcome in NSCLC Treated With EGFR Tyrosin Kinase Inhibitors (TKI)
Brief Title: Early Changes in Positron Emissions Tomography (PET/CT) Scan as Predictors of Clinical Outcome in NSCLC Treated With EGFR Tyrosin Kinase Inhibitors (TKI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thomas
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2014-01

CONDITIONS: Non-small Cell Lung Cancer Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-FDG-PET scan (Experimental): An early evaluation 18F-FDG-PET scan after 7-10 days
  Interventions: Procedure: 18F-FDG-PET scan

INTERVENTIONS:
Procedure: 18F-FDG-PET scan

SUMMARY:
Erlotinib, an anti-cancer agent targeting the epidermal growth factor receptor (EGFR), is an active treatment of patients with non-small cell lung cancer (NSCLC). Effect of treatment is primary seen in patients harboring a mutation in the EGFR. However, 10-15% of patients does not harbor a mutation but respond as well. Identifying these patients is a problem and methods are lacking.

Studies have shown that an early 18F FDG-PET might can predict response and outcome in these patients, but further studies are needed to confirm these findings.

ELIGIBILITY:
Inclusion Criteria:

* Lung Cancer patients with non-small cell histology and stage IV disease
* candidate for erlotinib treatment as first/ second/ third line of treatment

Exclusion Criteria:

* pregnancy
* severe dyspnoea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
18F-FDG-PET evaluation | Time to progression and latest april 2015 (up to 2 years)
  Standardized Uptake Values (SUV) will be used as measurement of 18F-FDG uptake

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Jylland, Denmark